CLINICAL TRIAL: NCT02361892
Title: The Effect of UPA on Women Ovarian Reserve
Brief Title: The Effect of Ulipristal Acetate (UPA) on Women Ovarian Reserve
Acronym: UPA_ovAge
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full professor, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPA and ovarian reserve
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
Keywords: ovarian reserve; infertility; leiomyomas; ulipristal acetate
MeSH Terms: conditions — Infertility; Leiomyoma | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulipristal acetate (Experimental): Women will be treated with 5mg/die of Ulipristal acetate for 2 courses of 3 months each
  Interventions: Drug: ulipristal acetate

INTERVENTIONS:
Drug: ulipristal acetate — 5 mg/day will be administered starting from day 1 of the cycle for two courses of 3 months each
  Other Names: Esmya

SUMMARY:
The uterine leiomyoma is the most common female benign disease.UPA seems to be most effective for the medical management of fibroids and could be place as preoperative adjunct to surgery but also as medical therapy to avoid surgery. No data have been published about the effect of UPA on FSH (Follicle stimulating hormone) or AMH levels nor on ovarian antral follicle count (AFC) or vascularization indexes during and after treatment. Considering that in young women of reproductive age (under 40 years old), desiring pregnancy, UPA has been proposed to avoid or postpone surgery, also in a long-term administration program, data about its effect on women ovarian reserve are urgently needed.

For these reasons, data on biochemical (AMH, FSH and E2) and 3D ultrasonographic (VI, Flow index, AFC) parameters of women treated by UP are needed to assess the effect of the drug in terms of ovarian reserve modification.

DETAILED DESCRIPTION:
The uterine leiomyoma is the most common benign tumor of the female genital tract. The myomas are usually clinically apparent in 25% of patients. Among the latest possible therapeutic options, UPA has proved to be most effective for the medical management of fibroids. Its advent in the clinical practice will probably modify the surgical approach, since UPA could possible place as a preoperative adjunct to surgery but also as medical therapy to avoid surgery. Very recently, the results of the first study on long-term intermittent (18 months) therapy with 10-mg UPA were published, demonstrating that this regimen (four courses of 3 months) maximizes the effect of UPA by inducing a very high rate of amenorrhea and reducing fibroid size.

Long term treatment, however, call in question safety issue that need to be explore. In patients treated by UPA, Estradiol under 5-mg and 10-mg doses remained at midfollicular levels after the first course of therapy, avoiding menopausal symptoms, as frequently observed in the gonadotropin-releasing hormone (GnRH-) agonist group. No data have been published about Estradiol levels at the end of second, third and fourth courses of UPA. Moreover, no data have been published about the effect of UPA on FSH or AMH levels nor on ovarian antral follicle count (AFC) or vascularization indexes during and after treatment. Considering that in young women of reproductive age (under 40 years old), desiring pregnancy, UPA has been proposed to avoid or postpone surgery, also in a long-term administration program, data about its effect on women ovarian reserve are urgently needed.

For these reasons, data on biochemical (AMH, FSH and E2) and 3D ultrasonographic (VI, FI, AFC) parameters of women treated by UP are needed to assess the effect of the drug in terms of ovarian reserve modification.

ELIGIBILITY:
Inclusion Criteria:

* submucosal,
* intramural or subserosal leiomyomas,
* symptoms of menometrorrhagia,
* menstrual disorder,
* infertility,
* pelvic pain

Exclusion Criteria:

* endometrial hyperplasia with atypia,
* estrogen-progestin therapy in the 2 months before enrollment,
* autoimmune diseases,
* chronic, metabolic, systemic and endocrine disorders, including hyperandrogenism, hyperprolactinemia, diabetes mellitus and thyroid disease,
* hypogonadotropic hypogonadism,
* majors clinical conditions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ovarian age change after two courses of UPA | In the follicular phase of the month before treatment and during the fifth month of treatment
  Ovarian Age will be assessed as a composite outcome by measuring FSH, Estradiol, AMH, 3D-AFC, VI, FI and VFI (vascularization flow index) in the follicular phase of the menstrual cycle before the start of treatment. The assessment will be repeated during the fifth month of UPA assumption. change will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD,PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Catanzaro, Italy